CLINICAL TRIAL: NCT03480295
Title: Exploring the Effects of a Preservative-free Ophthalmic Solution Containing Hyaluronic Acid 0.4% and Taurine 0.5% on the Ocular Surface of Glaucoma Patients Under Multiple Long-term Topical Hypotensive Therapy
Brief Title: Effects of a PF Ophthalmic Solution Containing HA0.4% and TAU 0.5%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRCCS-Fondazione GB Bietti
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA0.4%+TAU0.5% (Experimental): Patients had to administer 4 drops/day of an ophthalmic solution containing hyaluronic acid 0.4% and taurine 0.5% in addition to the ongoing glaucoma treatment
  Interventions: Device: Hyaluronic acid 0.4% and Taurine 0.5%
- HA0.2% (Active Comparator): Patients took 4 drops/day of an ophthalmic solution containing hyaluronic acid 0.2%
  Interventions: Device: Hyaluronic acid 0.2%

INTERVENTIONS:
Device: Hyaluronic acid 0.4% and Taurine 0.5% — 4 drops /day in addition to the ongoing glaucoma treatment
  Arms: HA0.4%+TAU0.5%
Device: Hyaluronic acid 0.2% — 4 drops /day in addition to the ongoing glaucoma treatment
  Arms: HA0.2%

SUMMARY:
Eligible patients underwent evaluation of ocular surface parameters by Ocular Surface Disease Index (OSDI) and Glaucoma Symptom Scale (GSS) questionnaires, Break Up Time test (BUT), Schirmer I test, corneal and conjunctival staining (Oxford scale) and conjunctival in vivo confocal microscopy (Heidelberg Retina Tomograph 3, Heidelberg Engineering Gmbh, Heidelberg, Germany). After the baseline visit, patients were randomized to use a PF ophthalmic solution containing HA 0.4% and TAU 0.5%, QID, in both eyes (Group 1) or to use a PF ophthalmic solution containing HA 0.2%, QID, (Group 2) in addition to the ongoing preserved hypotensive treatment. Follow-up visits were scheduled at 30 and 90 days.

DETAILED DESCRIPTION:
At the screening visit all patients underwent comprehensive ophthalmological examination including best corrected visual acuity assessment, slit lamp evaluation, IOP measurement using Goldmann applanation tonometry, and indirect dilated ophthalmoscopy with a 90 diopters lens. Visual field testing using Humphrey 24-2 SITA-Standard program (Carl Zeiss Meditec, Inc., Dublin, CA 24-2 program) was performed only for those patients with the last exam older than 3 months.

Baseline visit was splitted in two visits scheduled 1 week apart 2 days, to evaluate ocular surface alterations by means of several tests.

To minimize the influence of each test on the subsequent test, we performed first the least invasive and then the most invasive test. During the first baseline visit patients were asked to fill two questionnaires, the Ocular Surface Disease Index (OSDI) and the Glaucoma Symptom Scale (GSS) and then underwent the Break Up Time test (BUT), corneal and conjunctival staining evaluation using Oxford Staining Scheme, and Schirmer I test after 15 minutes of rest. During the second baseline visit, patients underwent conjunctival Confocal Laser Microscopy with the Rostock Module of Cornea of the Heidelberg Retina Tomograph (HRT3, Heidelberg Engineering Gmbh, Heidelberg, Germany).

At the end of the second baseline visit patients were randomized in two groups with a 1:1 ratio according to a computer-generated randomization list.

Group 1 (HA0.4%+TAU0.5%) was asked to self-administer 1 drop four times/day of a preservative-free ophthalmic solution containing 750KDa HA 0.4% and TAU 0.5% in both eyes, while Group 2 (HA0.2%) was asked to self-administer 1 drop four times/day of a preservative-free ophthalmic solution containing only 750KDa HA 0.2%, in addition to the ongoing hypotensive therapy.

Follow-up visits were scheduled at 30 and 90 days and all the exams were repeated in the same order, as they were performed at the baseline visits.

Both eyes were tested but only one randomly selected eye per patient was included in the analysis.

The primary endpoint was the comparison of the changes over time of the CGC density between the two groups. Secondary endpoints were the between groups comparisons of the changes over time of BUT, Schirmer test, conjunctival staining, OSDI score and GSS score.

All clinical measurements as well the statistical analysis were performed by investigators masked for the patients' treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma with an ongoing topical therapy with two or more preserved ocular hypotensive eye-drops per day for at least two years.

Exclusion Criteria:

* Best corrected visual acuity ≤ 20/40
* History of active or past ophthalmological diseases different than glaucoma
* Contraindications to use of topical solution components used in this study
* Current use of contact lenses
* Current use or use in the past 6 months of ocular medications other than hypotensive eye-drops
* Systemic treatments known to affect tear secretion
* Any history or slit lamp evidence of eye surface diseases different from dry eye
* History of ocular trauma
* Surgery or laser treatments
* Rheumatologic and autoimmune diseases
* Diabetes
* Peripheral neuropathies
* Use of systemic steroids or immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline of conjunctival goblet cells (CGC) density after 30 and 90 days | Baseline, 30 and 60 days
  Density of CGC was measured by means of conjunctival confocal microscopy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberti G, Agnifili L, Berardo F, Riva I, Figus M, Manni G, Quaranta L, Oddone F. Prospective, Randomized, Single Masked, Parallel Study Exploring the Effects of a Preservative-Free Ophthalmic Solution Containing Hyaluronic Acid 0.4% and Taurine 0.5% on the Ocular Surface of Glaucoma Patients Under Multiple Long-Term Topical Hypotensive Therapy. Adv Ther. 2018 May;35(5):686-696. doi: 10.1007/s12325-018-0699-8. Epub 2018 Apr 23. PMID 29687335